CLINICAL TRIAL: NCT03417401
Title: Phase Ib Study on Surgical Stabilizer Assisted Retinal Vein Cannulation (RVC) With tPA Infusion Confirmed by Intraoperative Angio-optical Coherence Tomography (Angio-OCT) for the Treatment of Central Retinal Vein Occlusion (CRVO).
Brief Title: Surgical Stabilizer Assisted RVC With rtPA for CRVO
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: organizationally not yet possible
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S61283
Record Dates: First submitted 2017-11-20; First posted 2018-01-31 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Central Retinal Vein Occlusion
MeSH Terms: conditions — Retinal Vein Occlusion | interventions — Vitrectomy; Tissue Plasminogen Activator; Infusions, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- RVC with tPA for CRVO (Experimental): Single arm phase I open label study were CRVO patients will have a vitrectomy with retinal vein cannulation and a single infusion of tPA (0.25mg/ml) intravenously with a maximum dose of 1mg.
  Interventions: Procedure: Vitrectomy with retinal vein cannulation and intravenous rtPA (Actilyse) infusion up to 1mg.; Drug: Intravenous Infusion

INTERVENTIONS:
Procedure: Vitrectomy with retinal vein cannulation and intravenous rtPA (Actilyse) infusion up to 1mg. — Standard 3-port pars plana vitrectomy with surgical stabilizer assisted ( surgical robot) retinal vein cannulation with recombinant tissue Plasminogen Activator (Actilyse-0.25mg/ml) infusion with a maximal dose of 1mg..
Drug: Intravenous Infusion — Intravenous infusion in a retinal vein with rtPA (Actilyse 0.25mg/ml).
  Other Names: Recombinant tissue Plasminogen Activator (rtPA)

SUMMARY:
This phase Ib study investigates the safety and efficacy of performing a retinal vein cannulation with recombinant tissue Plasminogen Activator infusion into a retinal vein with the help of an updated dedicated surgical stabiliser for the treatment of central retinal vein occlusion.

DETAILED DESCRIPTION:
Investigator-initiated, unmasked, single-arm, mono-center, prospective, interventional case series phase Ib trial. In line with the previous phase I trial, this trial will be biphasic; first 3 patients will be included, when the procedure and product prove to be safe and an added value is noted from the intra-operative OCT-angiography, another 3 will be included afterwards (≥21 days between last inclusion of the first group and first inclusion of the second group).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years
* Recent diagnosis (<8 weeks) of CRVO
* Recent onset of symptoms (<12 weeks)
* Visual acuity < 5/10 in study eye
* Visual acuity >1/10 in fellow eye
* Central macular thickness >250µm
* Signed informed consent prior to inclusion

Exclusion Criteria:

* Fluorescein allergy
* Active neovascularization
* Eye disease other than CRVO or Cataract decreasing central vision
* History of retinal surgery
* High myopia (> -10D)
* Contraindication for the use of systemic anticoagulant medication
* Extensive macular ischemia noted on fluo-angiography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10-16 (Estimated); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Success rate of retinal vein cannulation | 10 min
  successful cannulation defined as peroperatively seen washout of blood in the cannulated retinal vein. The success rate is defined as the number of successful cannulations divided by the total number of cannulation attempts.
number of intervention-related surgical complications | 7 days
  These exist of the intra-operative occurence of:
  * retinal vein tear (visually seen by the surgeon)
  * uncontrollable vitreous cavity hemorrhage (as seen by the surgeon)
  * retinal tear in the proximity of the cannulation site (as seen by the surgeon)
  * intra-/subretinal injection (as seen by the surgeon)
  * breakage of the needle (as seen by the surgeon)
  * failure of stabilizer in holding the instrument immobilized in a certain position (as seen by the surgeon)
duration of infusion | 10 minutes
  The time of infusion measured during surgery with a maximum of 10 minutes
number of intervention-related non-surgical complications | 7 days
  The postoperative occurence of:
  * hemorrhagic cerebrovascular accidents due to rtPA (confirmed by CT-scan and neurological examination after referral to the neurologist)
  * large hemorrhage elsewhere to be related with the use of rtPA (as confirmed by clinical examination and/or CT-scan/ultrasound after referral to vascular surgeon)

SECONDARY OUTCOMES:
change in visual acuity after 6 to 8 weeks | 6-8 weeks
  best corrected visual acuity tested with ETDRS chart
change in central macular thickness after 6 to 8 weeks | 6-8 weeks
  measurement of central macular thickness with spectral domain-OCT
intra-/postoperative complications not related to the surgical stabilizer / retinal vein cannulation / rtPA | 7 days
  - complications of intraocular surgery:
  * wound leak tested with concentrated fluorescein (Seidel effect present/absent)
  * endophthalmitis as seen with the slit lamp/ultrasonography
  * post-operative macular edema objectivated with OCT imaging
  * vitreous hemorrhage > 2 weeks after intervention as seen at the slit lamp and confirmed with ultrasonography
  * development of neovascularization as seen at the slit lamp / fluorescein angiogram
intra-/postoperative complications not related to the surgical stabilizer / retinal vein cannulation / rtPA | 7 days
  - complications during cataract surgery:
  * iris hemorrhage as seen through the surgical microscope (present/absent)
  * choroidal swelling as seen through the surgical microscope (present/absent)
  * suprachoroidal hemorrhage as seen through the surgical microscope (present/absent)
  * capsule tear as seen through the surgical microscope (present/absent)
  * dropped lens/intraocular lens (IOL). Recombinant tissue Plasminogen Activator (rtPA) as seen through the surgical microscope (occurred/not occurred)
intra-/postoperative complications not related to the surgical stabilizer / retinal vein cannulation / rtPA | 7 days
  - complications during vitrectomy:
  * retinal tears as seen through the surgical microscope (occurred/not occurred)
  * vitreous hemorrhage as seen through the surgical microscope (occurred/not occurred)
  * choroidal swelling as seen through the surgical microscope (present/absent)
  * suprachoroidal hemorrhage as seen through the surgical microscope (present/absent)
change in retinal flow intraoperatively visualized with OCT-angiography | 1 hour
  OCT-angiography visualized flow inside the retinal veins with the intraoperative OCT device; if there is flow the blood vessel is imaged in bright white, if there is no flow the blood vessel is not visible with angio-OCT.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Stalmans, Principal Investigator — UZ Leuven
Locations (1):
- Universitaire Ziekenhuizen Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No